CLINICAL TRIAL: NCT00925990
Title: A Trial of CTS-1027 in Interferon-Naive Hepatitis C Patients
Brief Title: CTS-1027 in Interferon-Naive Hepatitis C Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTS-1027-03
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Results first posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-02

CONDITIONS: Hepatitis C
Keywords: HCV; interferon-naive
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CTS-1027 + ribavirin (Experimental): Study drug plus ribavirin
  Interventions: Drug: ribavirin; Drug: CTS-1027
- CTS-1027 + placebo (Experimental): Study drug plus placebo for ribavirin
  Interventions: Drug: CTS-1027; Drug: Placebo for ribavirin

INTERVENTIONS:
Drug: ribavirin — 200 mg capsules, either 1000 or 1200 mg taken twice daily for up to 24 weeks
  Other Names: Copegus
  Arms: CTS-1027 + ribavirin
Drug: CTS-1027 — 5 and 10 mg tablets, 15 mg taken twice daily, for up to 24 weeks
Drug: Placebo for ribavirin — Capsules identical to ribavirin in appearance containing inactive ingredients
  Arms: CTS-1027 + placebo

SUMMARY:
The study is intended to determine whether CTS-1027 either alone or in combination with ribavirin is safe and effective in Hepatitis C patients who have not previously been treated with interferon.

DETAILED DESCRIPTION:
There are approximately 1 million Hepatitis C (HCV) patients in the US who have failed to respond to, or cannot tolerate, interferon or interferon plus ribavirin therapy. Significant adverse effects of interferon therapy include bone marrow depression (with reduced white blood cell and platelet counts) and major psychiatric disorders (especially depression). Ribavirin is associated with hemolytic anemia in a minority of patients who are treated with it. Patients with chronic HCV infection have a very low incidence of spontaneous viral clearance, have progressive disease, and have a continuing medical need for more efficacious and safer therapy. There is a significant unmet medical need for therapy in HCV patients who cannot (or will not) tolerate interferon-based treatment.

This trial will evaluate the effects of CTS-1027 with or without ribavirin in patients who are previously untreated with interferon including patients with major psychiatric disorders, uncontrolled autoimmune disease, and patients who simply decline treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of minimum adult legal age (according to local laws for signing the informed consent document), able to provide written informed consent, and understand and comply with the requirements of the trial
* A history of chronic (> 6 months duration) genotype 1 Hepatitis C (HCV) infection
* Unsuitable for interferon-based HCV treatment, defined as at least one of the following three criteria:

  * Contra-indicated for interferon treatment due to current or prior psychiatric disorders
  * Patient's decision to not pursue interferon-based therapy
  * In the opinion of the Principal Investigator, the patient is not a suitable candidate for interferon-based therapy
* a-fetoprotein (AFP) <= 50 ng/mL
* Hemoglobin ≥ 12 g/dL, platelet count ≥ 100 x 109/L, and white blood cell count ≥ 1.5 x 109/L
* Willingness to utilize two reliable forms of contraception (for both males and females of childbearing potential) from screening to at least six months after the completion of the trial.

Exclusion Criteria:

* Decompensated or severe liver disease defined by one or more of the following criteria:

  * Prothrombin time 3 seconds > control
  * Direct bilirubin ≥ 1.5 x upper limit of normal range (ULN)
  * Serum albumin below normal limits
  * AST or ALT > 7 x ULN at screening
  * Evidence of portal hypertension including:

    1. Varices on esophagogastroduodenoscopy (EGD) with or without a history of gastrointestinal bleeding; or
    2. Ascites
* Cirrhosis defined by one or both of the following criteria:

  * Liver biopsy showing cirrhosis
  * Other clinical signs and symptoms suggestive of cirrhosis
* Prior therapy for HCV with an interferon-based regimen
* Hepatocellular carcinoma (HCC) or suspicion of HCC clinically or on ultrasound (or other imaging techniques)
* Known history or presence of human immunodeficiency virus (HIV) infection
* Co-infection with hepatitis B virus (HBV)
* If female: pregnant, lactating, or positive serum pregnancy test
* Renal impairment (creatinine > 1.5 x ULN), creatinine clearance < 50 mL/min, or hepatorenal syndrome
* Hospitalization for liver disease within 60 days of screening
* Use of concomitant or prior drug therapy for HCV three months prior to screening
* Use of drugs of abuse in the prior three months (allowed if medically prescribed or indicated)
* History of alcohol abuse (> 50 g per day) within the past year
* History or presence of clinically concerning cardiac arrhythmias or prolongation of pre-dose QT or QTc interval of > 450 milliseconds
* Other concomitant disease or condition likely to significantly decrease life expectancy (e.g., moderate to severe congestive heart failure) or any malignancy other than curatively treated skin cancer (basal cell or squamous cell carcinomas), unless adequately treated or in complete remission for ten or more years
* Any patient who has received any investigational drug or device within 30 days of dosing, or who is scheduled to receive another investigational drug or device during the course of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Castelloe, MD, Study Chair — Conatus Pharmaceuticals Inc.
Locations (21):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Medical Associates Research Group, San Diego, California
  - Kaiser Permanante, San Diego, California
  - VA Medical Center, San Diego, San Diego, California
  - University of Colorado Health Science Center, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainsville, Florida
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of MA Mem Med Ctr, Worchester, Massachusetts
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - MN Clinical Research Center, Plymouth, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - St. Louis University, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - University of NC at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Consultants of Clinical Research, Ohio GI and Liver Institute, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - VA Medical Center, Houston, Houston, Texas
  - VCU-Medical College of Virginia, Richmond, Virginia
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- CTS-1027 + Ribavirin: CTS-1027, 5mg and 10 mg tablets (one each) taken twice daily for a total daily dose of 30 mg.
  Ribavirin, 200 mg capsules, taken in two divided daily doses totaling 1000 mg daily for patients weighing 75kg or less, and 1200 mg daily for patients weighing more than 75 kg
- CTS-1027 + Placebo: CTS-1027, 5mg and 10 mg tablets (one each) taken twice daily for a total daily dose of 30 mg.
  Placebo, incactive capsules identical in appearance to ribavirin capusules. Five (for patients weighing 75 kg or less) or six (for patients weighing more than 75 kg) capsules taken in two divided daily doses.
Period: Overall Study
Arm/Group | CTS-1027 + Ribavirin | CTS-1027 + Placebo
Started | 35 | 35
Completed | 30 | 24
Not Completed | 5 | 11
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 1 | 1
Not completed — moved out of state, missed medication | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CTS-1027 + Ribavirin | CTS-1027 + Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 35 | 68
  >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 52.6 (6.8) | 49.7 (9.1) | 51.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 23 | 26 | 49
Region of Enrollment [Number; unit: participants]
  United States | 34 | 31 | 65
  Puerto Rico | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in HCV-RNA (Hepatitis C Virus Ribonucleic Acid) Levels From Baseline Through 24 Weeks of Treatment
Description: Measure the mean absolute changes in HCV-RNA (Hepatitis C virus ribonucleic acid, also known as "viral load") levels in the blood from before treatment (baseline) through 24 weeks of treatment.
  Mean Absolute Change in HCV-RNA (log) = log10(HCV-RNA Week 24) - log10(HCV-RNA Baseline)
Time Frame: Baseline and 24 weeks
Population: All patients receiving at least one dose of study drug were analyzed for safety.
Measure: Mean (Standard Deviation); unit: log (IU/mL)
Groups:
- CTS-1027 + Ribavirin: CTS-1027, 5mg and 10 mg tablets (one each) taken twice daily for a total daily dose of 30 mg.
  Ribavirin, 200 mg capsules, taken in two divided daily doses totaling 1000 mg (5 capsules) daily for patients weighing 75kg or less, and 1200 mg (6 capsules) daily for patients weighing more than 75 kg
Arm/Group | CTS-1027 + Ribavirin | CTS-1027 + Placebo
Number analyzed (Participants) | 35 | 35
log (IU/mL) | -0.48 (0.50) | -0.12 (0.76)

2. Secondary Outcome: Mean Change in Aminotransferases From Baseline to 24 Weeks of Treatment
Description: Mean absolute changes in ALT (alanine aminotransferase)in the blood from before treatment (baseline)through 24 weeks of treatment are presented.
  Mean absolute change in ALT (IU/ml)= ALT(Week 24) - ALT(baseline)
Time Frame: Baseline and 24 weeks
Population: All patients dosed with at least one dose of study drug were analyzed.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | CTS-1027 + Ribavirin | CTS-1027 + Placebo
Number analyzed (Participants) | 35 | 35
IU/mL | -15.6 (42.9) | -16.5 (65.5)

ADVERSE EVENTS:
Arm/Group | CTS-1027 + Ribavirin | CTS-1027 + Placebo
Serious Adverse Events (participants affected / at risk) | 3/35 | 6/35
Other Adverse Events (participants affected / at risk) | 31/35 | 29/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTS-1027 + Ribavirin (N=35) | CTS-1027 + Placebo (N=35)
colitis ulcerative (Gastrointestinal disorders) | 1 (2) | 0 (0)
lobar pneumonia (Infections and infestations) | 1 (2) | 0 (0)
spondylitic myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
staphylococcal abscess (Infections and infestations) | 0 (0) | 1 (1)
chest pain (General disorders) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
upper GI hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTS-1027 + Ribavirin (N=35) | CTS-1027 + Placebo (N=35)
anemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
vomiting (Gastrointestinal disorders) | 3 (5) | 1 (1)
diarrhea (Gastrointestinal disorders) | 3 (4) | 1 (2)
constipation (Gastrointestinal disorders) | 2 (3) | 1 (1)
fatigue (General disorders) | 11 (12) | 8 (8)
edema peripheral (General disorders) | 2 (2) | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3)
myalgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (4)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3)
dizziness (Nervous system disorders) | 2 (2) | 2 (2)
insomnia (Psychiatric disorders) | 5 (6) | 0 (0)
headache (Nervous system disorders) | 5 (6) | 5 (5)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 12 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less